CLINICAL TRIAL: NCT03679975
Title: A Single Center Study to Evaluate the Effect of Riluzole Oral Soluble Film on Swallowing Safety in Individuals With Amyotrophic Lateral Sclerosis
Brief Title: Riluzole Oral Soluble Film (ROSF) Swallowing Safety in Amyotrophic Lateral Sclerosis (ALS)
Acronym: ROSF
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The study is no longer required
Sponsor: Aquestive Therapeutics (Industry)
Collaborators: inVentiv Health Clinical (Other); Covance (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 17MO1R-0012
Record Dates: First submitted 2018-09-19; First posted 2018-09-21 (Actual); Results first posted 2020-08-10 (Actual); Last update posted 2020-08-18 (Actual); Status verified 2020-08

CONDITIONS: Amyotrophic Lateral Sclerosis
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis

STUDY DESIGN:
Intervention Model Description: The original plan was to enroll 30 patients for a final sample size of 25 completed patients. With agreement from the FDA, the Sponsor decided to terminate the study after 9 completed patients, based on an interim analysis of the first 8 completed patients with no evidence of a harmful effect of one dose of 50 mg Riluzole Oral Film on swallowing function.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Subjects with ALS (Experimental): Subjects with a diagnosis of probable or definite ALS in accordance with the Revised El-Escorial Criteria were administered a single dose of the Riluzole Oral Soluble Film (ROSF) 50 mg.
  Interventions: Drug: Riluzole Oral Soluble film (ROSF) 50 mg

INTERVENTIONS:
Drug: Riluzole Oral Soluble film (ROSF) 50 mg — Enrolled subjects underwent an instrumental evaluation of swallowing safety before and after administration of a single dose of the ROSF formulation containing 50 mg of riluzole.
  Other Names: ROSF; Riluzole Orodispersible Film (ROF)

SUMMARY:
The primary objective is to evaluate the effect, if any, of a single 50 mg dose of Riluzole Oral Soluble Film (ROSF) on swallowing safety in individuals with amyotrophic lateral sclerosis.

DETAILED DESCRIPTION:
This was a single site, single dose, open-label study with one group of male or female patients between 18-80 years old with a diagnosis of Probable or Definite Amyotrophic Lateral Sclerosis (ALS) according to revised El-Escorial Criteria. Patients seen in the ALS Clinic at the University of Florida were screened to determine eligibility for participation in the study according to the specified inclusion/exclusion criteria. Following informed consent and enrollment, subjects were given a complete physical and neurological examination including the validated Amyotrophic Lateral Sclerosis Functional Rating Scale-Revised (ALSFRS-R). Swallowing safety was assessed using the gold standard Videofluoroscopic Swallowing Study (VFSS) to allow direct visualization of the swallowing process and any episodes of penetration or aspiration were quantified using the validated Penetration Aspiration Scale (PAS). Subjects participated in a standardized protocol that includes 11 bolus stimuli presentations of different liquid and food materials to test swallowing function using a progression of textures and materials. Immediately following this assessment, subjects were given a single dose of ROSF 50 mg, placed on the median lingual sulcus of the dorsum of the tongue (area under the tongue on the midline groove that separates the surface of the tongue into right and left halves). Three minutes after the administration of ROSF, the identical standardized VFSS protocol was re-administered to allow a comparison of swallowing safety (using the PAS scale) pre- versus post-ROSF administration.

The original plan was to enroll 30 patients for a final sample size of 25 completed patients. The protocol stipulated that, depending upon the study enrollment rate, the Sponsor could elect to perform an interim analysis using available data from the subset of subjects who had completed the study at that time. An interim assessment of the data was performed after 8 subjects had completed the study and a ninth patient had been screened and was awaiting VFSS. With agreement from the FDA, the Sponsor decided to terminate the study after 9 completed patients, based on the analysis of the first 8 completed patients showing no evidence of a harmful effect of one dose of ROSF 50 mg on swallowing function.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects between 18-80 years of age, inclusive
2. Subjects with a diagnosis of probable or definite ALS in accordance with the Revised El-Escorial Criteria
3. Subjects must be currently on an oral diet and able to take foods and liquids by mouth equivalent to a score of 3 or above on the Functional Oral Intake Scale.
4. Subjects with no known allergy to barium, riluzole or inactive ingredients in ROSF
5. Subject or subject's legally authorized representative must be willing and able to give informed consent/assent and HIPAA authorization.
6. Subject must have the ability to comprehend and be informed of the nature of the study, as assessed by the Principal Investigator or Sub-Investigator.
7. Subjects prescribed riluzole at or before the dose of study drug. (The study was open to subjects currently taking riluzole at screening, subjects who were not currently taking riluzole at screening who had taken riluzole in the past, and subjects to be newly started on riluzole (given as ROSF in this study).
8. Availability to volunteer for the entire study duration and willing to adhere to all protocol requirements
9. Female subjects of childbearing potential (i.e. not surgically sterile, not 2 years postmenopausal, or not with a sterile partner) must have a negative pregnancy test at Screening and Visit 1, agree to abstinence, be practicing double barrier contraception or using an FDA approved barrier method contraceptive (e.g., licensed hormonal or barrier methods) for more than 2 months prior to the screening visit and commit to an acceptable form of birth control for the duration of the study and for 30 days after participation in the study.

Exclusion Criteria:

1. Subjects who score 2 or below on the Functional Oral Intake Scale.
2. Subjects with a prior swallowing study that has shown a Penetration Aspiration Scale score of 3 or greater
3. Subjects with a history of 2 or more episodes of aspiration pneumonia requiring hospitalization
4. Subjects with a history of clinically significant liver disease, renal disease, or any other medical condition judged to be exclusionary by the Investigator
5. Subjects who were unwilling to sign informed consent or subjects who for any other reason in the judgment of investigator were unable to complete the study
6. Female subjects who had a positive urine pregnancy test (βhCG) at screening or Visit 1, were trying to become pregnant, or were breastfeeding.
7. Subjects with active cancer within the previous 2 years, except treated basal cell carcinoma of the skin
8. Subjects who had taken any experimental drug within 30 days prior to enrollment or within 5 half-lives of the investigational drug -whichever was the longer period. However, subjects who had previously completed other Aquestive Therapeutics-sponsored ROSF clinical studies within the last 30 days prior to enrollment could be eligible for consideration for entry into this study.
9. Subjects with known history of moderate or severe renal impairment as defined by a calculated creatinine clearance of ≤50 mL/minute
10. Subjects currently taking riluzole with alanine aminotransferase levels greater than 5 times upper limit of normal or with evidence of clinical jaundice. (Riluzole should be discontinued in these patients.)
11. Subjects who would be receiving riluzole for the first time who exhibited baseline elevations of several liver function tests (especially elevated bilirubin). (These findings at baseline should preclude the use of riluzole including ROSF).
12. Use of potentially hepatotoxic drugs: (e.g., allopurinol, methyldopa, sulfasalazine).
13. Subjects with clinically significant abnormal laboratory values in the judgment of the Investigator
14. Use of strong or moderate CYP1A2 inhibitors (e.g., ciprofloxacin, enoxacin, fluvoxamine, methoxsalen, mexiletine, thiabendazole, vemurafenib, zileuton) and CYP1A2 inducers (e.g. rifampin and barbiturates) in the previous 30 days before first drug administration.
15. Anything else that, in the opinion of the Investigator, would place the subject at increased risk or preclude the subject's full compliance with or completion of the study.
16. Employee or immediate relative of an employee of the investigator, Aquestive Therapeutics, any of its affiliates or partners, or inVentiv Health.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2018-04-04 (Actual); Primary Completion 2018-09-26 (Actual); Study Completion 2018-12-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Cassie Jung, Study Director — Aquestive Therapeutics
Locations (1):
- University of Florida Center for Movement Disorders & Neuroscience, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Eleven subjects were screened for the study: Two subjects withdrew after signing informed consent but prior to any study procedure. Nine subjects were enrolled and received study medication and completed the study. There were no discontinuations.
Pre-assignment Details: Planned enrollment was 30 patients for a final sample size of 25 completed patients. The Sponsor decided to terminate the study after 9 completed patients (with agreement from the FDA), based on an interim analysis of the first 8 completed patients with no evidence of a harmful effect of 1 dose of 50 mg Riluzole Oral Film on swallowing function.
Groups:
- Patients With ALS With Single 50 mg Dose ROSF: Single group of patients with a diagnosis of probable or definite ALS in accordance with the Revised El-Escorial Criteria.
  They participated in a Videofluoroscopic Swallowing Study (VFSS) with 11 bolus trials and were scored by two independent raters on the Penetration Aspiration Scale (PAS). They were then given a single dose of 50 mg Riluzole Oral Film, and the Videofluoroscopic Swallowing Study was repeated at three minutes after dosing.
Period: Overall Study
Arm/Group | Patients With ALS With Single 50 mg Dose ROSF
Started | 9
Completed | 9
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Subjects With ALS: Subjects with a diagnosis of probable or definite ALS in accordance with the Revisited El-Escorial Criteria will be administered a single dose of the Riluzole Oral Soluble Film (ROSF) 50 mg.
  Riluzole Oral Soluble film (ROSF) 50 mg: Enrolled subjects will undergo an instrumental evaluation of swallowing safety before and after administration of a single dose of the ROSF formulation containing 50 mg of riluzole.
Arm/Group | Subjects With ALS
Number analyzed (Participants) | 9
Age, Continuous [Mean (Full Range); unit: years] | 61 [37 to 77]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 7
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 7
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 9
Change in Penetration Aspiration Scale Score on Videofluoroscopic Study before and after a single do [Count of Participants; unit: Participants] — Subjects participated in a Videofluoroscopic Swallowing Study (VFSS) with 11 bolus trials and were scored by two independent raters on the Penetration Aspiration Scale (PAS). They were then given a single dose of 50 mg Riluzole Oral Film, and the Videofluoroscopic Swallowing Study was repeated at three minutes after dosing. The primary outcome was change on PAS scores from pre- to post-dose.
  Participants | 5

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Categorized by Differences From Baseline in Penetration Aspiration Scale (PAS) - Sum of Scores Method
Description: Swallowing safety was assessed using the gold standard Videofluoroscopic Swallowing Study (VFSS) to allow direct visualization of the swallowing process and any episodes of penetration or aspiration were quantified using the validated Penetration Aspiration Scale (PAS). The PAS is an 8-point validated scale of swallowing safety that takes into account both degree/level of airway invasion during swallowing and the patients' response to the penetration or aspiration episode. The assessment is performed via videofluoroscope. Scores of 1 and 2 indicate airway safe swallowing with no airway invasion or ability to clear airway invasion. Scores 3 through 8 indicate airway unsafe swallowing based on penetration of the airway, level of penetration, and the patient's ability to respond. An increase in score/higher score means a worse outcome. A decrease in score/lower score means a better outcome.
Time Frame: Before and after administration of ROSF 50 mg on day 1 (visit 1)
Population: Safety Population comprising all enrolled subjects who received the single ROSF 50 mg administration.
Measure: Count of Participants; unit: Participants
Groups:
- Subjects With ALS: Subjects with a diagnosis of probable or definite ALS in accordance with the Revised El-Escorial Criteria will be administered a single dose of the Riluzole Oral Soluble Film (ROSF) 50 mg.
  Riluzole Oral Soluble film (ROSF) 50 mg: Enrolled subjects will undergo an instrumental evaluation of swallowing safety before and after administration of a single dose of the ROSF formulation containing 50 mg of riluzole.
Arm/Group | Subjects With ALS
Number analyzed (Participants) | 9
Participants
  Increase in sum of scores post dose | 0
  Same sum of scores post dose | 7
  Decrease in sum of scores post dose | 2

ADVERSE EVENTS:
Time Frame: From screening until 1 day post-dose
Arm/Group | Subjects With ALS
All-Cause Mortality (participants affected / at risk) | 0/9
Serious Adverse Events (participants affected / at risk) | 0/9
Other Adverse Events (participants affected / at risk) | 0/9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2017-10-18): https://cdn.clinicaltrials.gov/large-docs/75/NCT03679975/Prot_000.pdf
  • Statistical Analysis Plan (2018-10-12): https://cdn.clinicaltrials.gov/large-docs/75/NCT03679975/SAP_001.pdf